CLINICAL TRIAL: NCT03423953
Title: Comprehensive Nano Post Market Data Collection
Brief Title: Comprehensive Nano - Post Market Clinical Follow-Up Study
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.GE2.13
Record Dates: First submitted 2018-01-29; First posted 2018-02-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis; Revision; Correction of Functional Deformity
Keywords: osteoarthritis; avascular necrosis; rheumatoid arthritis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Anatomic: Patients receiving the Anatomic or Hemi verison of the Comprehensive Nano.
  Interventions: Device: Comprehensive Nano
- Reverse: Patients who have received the Reverse version of the Comprehensive Nano.
  Interventions: Device: Comprehensive Nano

INTERVENTIONS:
Device: Comprehensive Nano — Patients requiring the Comprehensive Nano shoulder system.

SUMMARY:
This data collection project is intended to provide clinical outcomes data to engineering, marketing as well as fulfill the post market surveillance requirements of various regulatory authorities. The study will be a prospective and one-arm.

DETAILED DESCRIPTION:
The Comprehensive® Shoulder System with Nano humeral component is a humeral prosthesis system intended for use in total or hemi shoulder arthroplasty surgery. Total shoulder arthroplasty consists of replacement of the humeral head and glenoid. Hemi-arthroplasty consists of replacement of only the humeral head.

This project is a prospective study including one-hundred and fifty (150) anatomic and hemi cases and 44 reverse shoulders collected from up to ten (10) sites. All potential study subjects will be required to participate in the Informed Consent process.

ELIGIBILITY:
Inclusion Criteria:

* Non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis.
* Rheumatoid arthritis
* Revision where other devices or treatments have failed
* Correction of functional deformity.
* Difficult clinical management problems where other methods of treatment may not be suitable or may be inadequate
* Difficult clinical management problems where other methods of treatment may not be suitable or may be inadequate

Exclusion Criteria:

* Infection
* Sepsis
* osteomyelitis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients in need of an uncemented shoulder arthroplasty and who meet all of the inclusion and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Estimated)
Dates: Start 2013-10-30 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Survivorship | 10 years
  Kaplan Meier method

SECONDARY OUTCOMES:
ASES Score (American Shoulder and Elbow Surgeons) | 10 years
  Improvement in this score from preop to 10 year follow-up. This score includes 2 scales: 1 scale for pain, from 0 to 10 where 0 stands for "no pain at all" and 10 for "pain as bad as it can be". The second scale is for the stability of the shoulder, from 0 to 10 (0 stands for "very stable" and 10 for "very unstable").
SANE Score (Single Assessment Numeric Evaluation) | 10 years
  Improvement in this score from preop to 10 year follow-up. This is a simple, single-question, patient-based shoulder function assessment tool: "How would you rate your shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?"
Constant-Murley Score | 10 years
  Improvement in this score from preop to 10 year follow-up. This is a 100-point score. Higher scores indicate a better outcome.
X-rays evaluated for radiolucencies, osteolysis, migration and subsidence | 10 years
  Standard evaluation performed on both humeral and glenoid components

CONTACTS AND LOCATIONS:
Overall Officials: Paola Vivoda, Study Director — Zimmer Biomet
Locations (5):
- Privatklinik Leech, Graz, Styria, Austria
- Kingston General Hospital, Kingston, Ontario, Canada
- South Korea (2):
  - Chonnam National University Hospital, Gwangju
  - Samsung Medical Centre, Seoul
- University of Liverpool, Liverpool, Merseyside, United Kingdom